CLINICAL TRIAL: NCT06405399
Title: Design, Implementation and Evaluation of the Guided Observer Role in Clinical Simulation. A Pilot Study
Brief Title: Design, Implementation and Evaluation of the Guided Observer Role in Clinical Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Simulación
Record Dates: First submitted 2024-05-06; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Anaphylactic Reaction
Keywords: simulation training;; undergraduated students
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded in their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided observed (Experimental): Students attended the simulated clinical experience as non-participant observers, but were supported by an observation rubric. Observation took place in situ, within the simulation laboratory itself, in an adjacent video-monitored room.
  Interventions: Other: Educational intervention. observation guide
- Control group: Participant (No Intervention): Students attended the simulated clinical experience directly as participants.

INTERVENTIONS:
Other: Educational intervention. observation guide — An observation checklist based on the Lasater Clinical Judgment Rubric (LCJR) was created and adapted to the simulated clinical experience in order to address the learning outcomes to be achieved by nursing students. This resulted in a list of forty items divided into four main groups: patient safety (8 items), communication and relationship with the patient (7 items), teamwork (7 items) and technical skills (18 items).
  Other Names: Observation guide
  Arms: Guided observed

SUMMARY:
The aim of this study is to assess the effectiveness of the guided observed role in a simulation learning programme for nursing students in acquiring the competence (knowledge, skills and attitudes) to care for patients affected by anaphylactic situations. This will be achieved by comparing the participants' simulation roles with the guided observed role.

The design was that of an exploratory randomised controlled trial. The variables employed to assess the efficacy of the intervention were competence and its associated attributes. These were measured using a ten-question multiple-choice test to assess knowledge; the simulation performance assessment using the Creighton Simulation Evaluation Instrument to assess skill; the learner's perception of the simulation's effectiveness in meeting their learning needs, through the Simulation Effectiveness Tool Modified (SET-M). Furthermore, the extent to which reflective thinking was achieved during the simulation was evaluated using the Self-Debriefing Reflection Rubric. Additionally, the students' perceptions of their role were assessed through seven open-ended questions.

DETAILED DESCRIPTION:
The study was a prospective, randomised, double-blind controlled trial conducted from October to November 2023 at a Nursing Faculty. The participants were fourth-year Bachelor of Science in Nursing students from a University in the North of Spain. A convenience sample of students from the nursing programme participated in the study. The recommended sample size was 40 participants per group, accounting for a 10% allowance for withdrawals, missing data, and lost follow-up.

Following their registration to participate in the study, 123 students were screened by the researchers to determine their eligibility. Prior to the commencement of the research, the students were informed about the objectives and the project and they signed the informed consent form. Upon arrival at the simulation centre to develop the simulated experience, participants completed the pre-test assessment and were randomly assigned to either the intervention group (57 students) or the control group (56 students) at a 1:1 ratio using a computer-generated assignment. Following the simulation experience, participants completed the post-test assessment and the various tools of the research.

During the study, two participants in the intervention group and one in the control group were excluded due to missing follow-up (refusal to continue in the research), and one student in the control group was removed by statistical analysis. In total, 99 participants were included in the data analysis. The students completed the sociodemographic information (age, gender, and previous experience in simulation experiences with anaphylactic situations) and the data on different variables via the online platform Google Form.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the 4rd year of nursing at the Faculty of Nursing of the University of Navarra and who voluntarily agree to participate in the study.

Exclusion Criteria:

* Students who had previously undergone a simulated clinical experience of managing an anaphylactic shock.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Knowledge | two months
  In order to gauge the comprehension of information pertaining to a case of anaphylactic shock, a questionnaire comprising 10 multiple-choice inquiries, each presenting four possible responses, was devised. This questionnaire encapsulates the primary algorithms delineating the contemporary approach to managing anaphylactic shock, as outlined by the European Resuscitation Council in 2021, alongside delineations of requisite nursing interventions.
Evaluation of the simulated experience: Creighton Simulation Evaluation Instrument (C-SEI) | Two month
  In order to assess the proficiency development of students allocated to the intervention group (guided observers) and the control group (participants), the Creighton Simulation Evaluation Instrument (CSEI) was employed. The CSEI, translated and validated into Spanish in 2019, comprises 22 dichotomous items divided into four different components: assessment, communication, critical creative, and technical skills. The Cronbach's alpha internal consistency coefficient for the entire scale was 0.839. The exclusion of any one of the questions was not found to significantly enhance the internal consistency of the scale.

SECONDARY OUTCOMES:
Self-Debriefing Reflection Rubric | Two months
  The tool comprised a set of six guiding questions, designed to assist with reflection on the experience based on Gibbs' (1988) Reflective Cycle. The questions are as follows: Q1-Description, Q2-Emotion, Q3-Evaluation, Q4-Analysis, Q5-Conclusion and Q6-Future Plan. The definitions of reflection levels proposed by Mezirow and the model of structured reflection were employed in the design of the Self-Debriefing Reflection Rubric for this study. The rubric comprised six items for the six questions, each with four possible rating levels. The responses were categorised as L-1 (Habitual Action), L-2 (Understanding), L-3 (Reflection), or L-4 (Critical Reflection). A mean rating of 3.0 or above for a student's submission indicated a consistent level of RT.
Simulation Effectiveness Tool - Modified (SET-M) | Two months
  In its updated form, the SET-M (Leighton, 2015) incorporates the simulation standards of best practices and terminology that have been established by the INACSL Standards Committee (INACSL Standards of Best Practice Simulation (INACSL Standards Committee, 2016)), The Quality and Safety Education for Nurses (QSEN) competencies (2007) and the Essentials of Baccalaureate Education for Professional Nursing Practice of the American Association of Colleges of Nursing (AACN) (2008). The SET-M is a useful instrument for evaluating the learner's perception of the effectiveness of the simulation in meeting their learning needs. The SET-M comprises 19 items, scored on a 3-point Likert scale: prebriefing (2 items), learning (6 items), confidence (6 items) and debriefing (5 items). The Spanish version of the SET-M was translated and validated, resulting in an internal consistency of 0.936 (Cronbach's alpha).
Open ended questions | Two months
  Seven open-ended questions were developed to ascertain the students' perceptions of their role (participant or guided observer) in the simulated clinical experience. A thematic review was conducted to identify the main categories, which were then used to inform the subsequent elaboration of the questions. For example, the question "Do you believe that the role of observer makes you more relaxed in the ECS?" was developed to assess the students' perceptions of the observer role. Similarly, the question "Has the observer role made you more passive in the ECS?" was designed to assess the students' views on the impact of the observer role on their behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Lizarbe Marta, PhD, Principal Investigator — University of Navarra Pamplona, Navarra, Spain
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain